CLINICAL TRIAL: NCT01884246
Title: Reducing Health Disparities in Appalachians With Multiple Cardiovascular Disease Risk Factors
Brief Title: Improving Heart Health in Appalachia
Acronym: HeartHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Moser (Other)
Collaborators: University of Kentucky Center for Excellence in Rural Health-Hazard (Unknown)
Responsible Party: Sponsor-Investigator, Debra Moser, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCORI 3048110484
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Hypertension; Hyperlipidemia; Depression
Keywords: lifestyle change; behavior change; obesity; hypertension; hyperlipidemia; physical inactivity; depression
MeSH Terms: conditions — Obesity; Hypertension; Hyperlipidemias; Depression; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-care CVD risk reduction (Experimental): A patient-centered, culturally appropriate lifestyle approach to promoting self-care in high risk patients.
  Interventions: Behavioral: Self-care CVD risk reduction; Other: Referral to primary care provider for CVD risk management
- Referral to primary care provider (Active Comparator): The study team provides a primary care provider for the patient, makes the referral and sends appropriate CVD risk reduction guidelines to the provider.
  Interventions: Other: Referral to primary care provider for CVD risk management

INTERVENTIONS:
Behavioral: Self-care CVD risk reduction — A patient-centered, culturally appropriate lifestyle approach to promoting self-care in high risk patients.
  Other Names: HeartHealth
  Arms: Self-care CVD risk reduction
Other: Referral to primary care provider for CVD risk management — The study team provides a primary care provider for the patient, makes the referral and sends appropriate CVD risk reduction guidelines to the provider.

SUMMARY:
Individuals in Appalachian Kentucky are vulnerable to cardiovascular disease (CVD) by virtue of having high rates of multiple CVD risk factors. There is a critical need to develop and test CVD risk reducing interventions that are appropriate and effective in Appalachia. In the absence of such interventions, the dramatic CVD disparities seen in this area will continue to rise.

Lifestyle interventions reduce CVD risk by 44%. The investigators and others have demonstrated that lifestyle change is most effective when patients are given the tools to engage in effective self-care, and that interventions individualized to patients' specific needs and barriers are more effective than interventions that are not. The central hypothesis is that to be successful in Appalachia, CVD risk reducing interventions must focus on patient-centered lifestyle change that increase individuals' abilities to engage in self-care, must be culturally appropriate, and must have components that overcome barriers faced by individuals living in Appalachia.

The investigators propose a randomized, controlled comparative effectiveness trial with 300 individuals from Appalachian Kentucky who do not have a primary care provider and who are at risk for CVD by virtue of having two or more modifiable CVD risk factors. The investigators will compare (1) a patient-centered, culturally appropriate, self-care CVD risk reduction intervention (HeartHealth) designed to improve multiple CVD risk factors while overcoming barriers to success with (2) referral of patients to a primary care provider for management of their CVD risk factors. The investigators propose the following specific aims to be tested at 4 months and 1 year after baseline. To compare the short and long-term impact of the interventions on:

1) the risk factor selected by patients (i.e., tobacco use, blood pressure, lipid profile, hemoglobin-A1c (HgA1c) for diabetics, body mass index, waist circumference, depressive symptoms, or physical activity level); 2) all of the CVD risk factors of each patient; 3) quality of life; 4) patient and healthcare provider satisfaction; 5) desirability and adoptability by assessing adherence to recommended CVD risk reduction measures, and retention of recruited individuals. The investigators hypothesize that in comparison to the referral strategy, the multifaceted patient-centered, self-care intervention will engender more favorable outcomes across all measures.

ELIGIBILITY:
Inclusion Criteria:

* residents of eastern Appalachian Kentucky
* do not have a primary care provider
* at risk for CVD as reflected by having two or more of the following modifiable risk factors

  1. clinical diagnosis of hypertension or taking medications diagnosed for hypertension or found to be hypertensive on screening;
  2. clinical diagnosis of hyperlipidemia or taking medication for treating abnormal lipid levels, or any lipid abnormality found on screening that indicates hyperlipidemia;
  3. diagnosis of type 2 diabetes or HgA1c > 7% found on screening;
  4. overweight or obese (body mass index ≥ 25 kg/m2);
  5. waist circumference > 40 inches in men or > 35 inches in women;
  6. clinical diagnosis of depression, on medications for depression or found to have depressive symptoms (score of > 9 on the Patient Health Questionnaire-9) by baseline screening;
  7. sedentary lifestyle meaning that the individual does not engage in at least 30 minutes of moderate activity for at least 4 days per week

Exclusion Criteria:

* known coronary artery disease, cerebrovascular disease, history of acute coronary syndrome or peripheral arterial disease;
* taking medications (e.g., protease inhibitors) that interfere with lipid metabolism;
* cognitive impairment that precludes an individual from understanding the consent process, answering questionnaires, or participating in the intervention;
* chronic drug abuse;
* end-stage renal or liver or pulmonary disease;
* current active cancer (i.e., undergoing active treatment for cancer) other than isolated skin cancer treatable by simple excision;
* gastrointestinal disease that requires special diets (e.g., Crohn's disease; celiac disease)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
cardiovascular risk factor selected by patient | 4 months
  Patient selects their own risk reduction goal from the following:
  smoking, blood pressure, lipid profile, body mass index, hemoglobin-A1c for diabetics, depression, physical activity level, waist circumference
cardiovascular risk factor selected by patient | 12 months
  Patient selects their own risk reduction goal from the following:
  smoking, blood pressure, lipid profile, body mass index, hemoglobin-A1c for diabetics, depression, physical activity level, waist circumference

SECONDARY OUTCOMES:
all CVD risk factors of each patient | 4 months
  All CVD risk factors that each patient has are secondary outcomes
all CVD risk factors of each patient | 12 months
  All CVD risk factors that each patient has are secondary outcomes

OTHER OUTCOMES:
quality of life | 4 months
quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Moser, DNSc, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States